CLINICAL TRIAL: NCT05168436
Title: Preferences Of Patients And Oncologists For The Characteristics Of The Treatment For RCC In Spain And Portugal
Brief Title: A Study of Preferences of Participants and Oncologists for the Characteristics of the Treatment for Renal Cell Carcinoma (RCC) In Spain And Portugal
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9W6
Record Dates: First submitted 2021-10-22; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Renal Cell Carcinoma
Keywords: OPDIVO®; Nivolumab; Preference; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with renal cell carcinoma (RCC) treated with nivolumab
- Cohort 2: Oncologists with expertise in renal cancer from Spain and Portugal

SUMMARY:
The purpose of this observational study is to determine patients' and professionals' preferences for the characteristics (attributes) of the treatment for Renal cell carcinoma (RCC) in Spain and Portugal.

DETAILED DESCRIPTION:
This study uses a literature review, qualitative (focus groups) and quantitative methods (discrete-choice experiment, DCE) to determine renal cell carcinoma (RCC) participants and oncologists' preferences. In this clinical trial, the study team will develop a survey consisting of comparisons of hypothetical treatment profiles (scenarios). Scenarios are presented to participants, and each participant chooses the most preferable.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Oncologists from Spain and Portugal will be identified by the promoter and invited to participate in the study in accordance with the inclusion criteria described below.

* The oncologist is currently working in a Spanish or Portuguese public hospital.
* The oncologist has at least 2 years of experience in the management of participants with Renal Cell Carcinoma (RCC).
* The oncologist has agreed to participate in the study.

Participants with a diagnosis of RCC will be identified and recruited by the Principal Investigators of the study, taking into account the inclusion criteria described below.

* The participant has been diagnosed with RCC for a minimum of 2 months before study inclusion.
* The participant has received or is currently receiving pharmacological treatment for RCC;
* The participant has provided the informed consent to participate in the study.
* The participant must be able to read, understand and complete the survey instrument according to the judgment of the responsible physician.

Exclusion Criteria:

• Not applicable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosis of Renal Cell Carcinoma (RCC) from a total of eight to eleven hospitals (6-8 located in Spain and 2-3 in Portugal) and oncologists with expertise in renal cancer from Spain and Portugal will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Utility: Renal cell carcinoma (RCC) participants' preferences | At Baseline
  Utility (preference score) derived for a treatment alternative choice (scenario)
Utility: Oncologists' preferences | At Baseline
  Utility (preference score) derived for a treatment alternative choice (scenario)

SECONDARY OUTCOMES:
Distribution of socio-demographic characteristics of Renal cell carcinoma (RCC) participants: Age | At Baseline
  Mean age, defined as the difference in time between date of birth and baseline visit
Distribution of clinical characteristics of RCC participants: Time since RCC diagnosis | At Baseline
  Mean time to diagnosis, defined as the differences in time between date of diagnosis and baseline visit
Distribution of socio-demographic characteristics of RCC participants: Place of residence | At Baseline
  Place of residence, defined as Province of residence categories at baseline visit
Distribution of socio-demographic characteristics of RCC participants: Gender | At Baseline
  Gender, defined as Gender categories at baseline visit, defined as female and male
Distribution of socio-demographic characteristics of RCC participants: Economic status (income) | At Baseline
  Economic status, defined as Euros per month
Distribution of socio-demographic characteristics of RCC participants: Education level | At Baseline
  Education level, defined as education level categories at baseline visit, defined as primary education, secondary education, university education, third-level studies (masters, doctorate, etc.)
Distribution of socio-demographic characteristics of RCC participants: Working situation | At Baseline
  Working situation, defined as working situation categories at baseline visit defined as full-time employed, part-time employed, self-employed, employed but on temporary sick leave due to RCC, permanent sick leave due to RCC, student, unemployed, retired, housework
Distribution of socio-demographic characteristics of RCC participants: Transport to the hospital: means, duration and cost | At Baseline
Distribution of socio-demographic characteristics of RCC participants: Other costs derived from the visit to the hospital (parking, meals...) | At Baseline
Distribution of clinical characteristics of RCC participants: American Joint Committee on Cancer (AJCC) Staging | At Baseline
  AJCC staging, defined as AJCC disease staging categories at baseline visit defined as Localized disease: Stages I and II; or advanced disease: Stages III and IV
Distribution of clinical characteristics of RCC participants: Charlson index | At Baseline
  Charlson index, defined as Mean score according to Charlson comorbidity index
Distribution of clinical characteristics of RCC participants: Karnofsky Performance Scale Index | At Baseline
  Karnofsky Performance Scale Index categories at baseline visit, defined as (0-100%); Lower score representing worst functional impairment
Distribution of clinical characteristics of RCC participants: Current drug treatment (if applicable) | At Baseline
  Current drug treatment, defined as drug treatment categories at baseline visit
Distribution of clinical characteristics of RCC participants: Identification of previous pharmacological treatments received by the participant for the treatment of RCC | At Baseline
  Previous drug treatment, defined as drug treatment categories at baseline visit
Distribution of clinical characteristics of RCC participants: Description of previous pharmacological treatments received by the participant for the treatment of RCC | At Baseline
  Previous drug treatment, defined as drug treatment categories at baseline visit
Distribution of socio-demographic characteristics of oncologists: Gender | At Baseline
  Gender, defined as Gender categories at baseline visit, defined as female and male
Distribution of socio-demographic characteristics of oncologists: Age | At Baseline
  Mean age, defined as the difference in time between date of birth and baseline visit
Distribution of socio-demographic characteristics of oncologists: Province where employed | At Baseline
  Province where employed, defined as Province categories at baseline visit
Distribution of socio-demographic characteristics of oncologists: Years of experience in RCC | At Baseline
  Years of experience in RCC, defined as Mean time of experience in RCC at baseline visit
Distribution of socio-demographic characteristics of oncologists: Years of experience in oncology | At Baseline
  Years of experience in oncology, defined as Mean time of experience in oncology at baseline visit
Distribution of socio-demographic characteristics of oncologists: Number of participants with RCC seen per year | At Baseline
  Number of participants with RCC seen per year, defined as Mean time of participants with RCC seen per year
Distribution of socio-demographic characteristics of oncologists: Other types of cancer treated | At Baseline
  Other types of cancer treated, defined as other cancers treated
Distribution of socio-demographic characteristics of oncologists: Level/ classification of hospital where employed | At Baseline
  Hospital level or classification categories at baseline visit, defined as first, second, third, and fourth level

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Castellon, Spain

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm